CLINICAL TRIAL: NCT02876835
Title: A Phase 3 Randomized, Open-label (Sponsor-blind), Active-controlled, Parallel-group, Multi-center, Event Driven Study in Non-dialysis Subjects With Anemia Associated With Chronic Kidney Disease to Evaluate the Safety and Efficacy of Daprodustat Compared to Darbepoetin Alfa
Brief Title: Anemia Studies in Chronic Kidney Disease: Erythropoiesis Via a Novel Prolyl Hydroxylase Inhibitor Daprodustat-Non-Dialysis (ASCEND-ND)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200808; 2016-000542-65 (EudraCT Number)
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Results first posted 2022-04-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Anaemia
Keywords: GSK1278863; hemoglobin; anemia; non-dialysis; erythropoiesis stimulating agents; daprodustat; chronic kidney disease
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Daprodustat (Experimental): Participants will receive oral daprodustat once daily.
  Interventions: Drug: Daprodustat; Drug: Placebo; Drug: Iron Therapy
- Darbepoetin alfa (Active Comparator): Participants will be administered darbepoetin alfa subcutaneously (SC).
  Interventions: Drug: Darbepoetin alfa; Drug: Placebo; Drug: Iron Therapy

INTERVENTIONS:
Drug: Daprodustat — The initial dose or oral daprodustat for ESA naïve subjects is based on Hgb and for ESA users is based on prior ESA dose. The dose is adjusted thereafter in order to achieve the target range.
  Arms: Daprodustat
Drug: Darbepoetin alfa — The initial dose of darbepoetin alfa to be administered for SC injection for ESA naïve subjects is based in Hgb and weight, and for ESA users is based on converting the prior ESA dose to the nearest available study darbepoetin alfa dose. The dose is adjusted thereafter in order to achieve the target range. IV darbepoetin alfa can be considered for participants transitioning to hemodialysis.
  Arms: Darbepoetin alfa
Drug: Placebo — Oral placebo tablets will be taken from Week -4 up to randomization (Day 1).
Drug: Iron Therapy — Participants will receive supplemental iron therapy if ferritin is <=100 ng/mL or TSAT is <=20%. The investigator will choose the route of administration and dose of iron.

SUMMARY:
The purpose of this multi-center event-driven study in non-dialysis (ND) participants with anemia associated with chronic kidney disease (CKD) is to evaluate the safety and efficacy of daprodustat compared to darbepoetin alfa.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 99 years of age (inclusive)
* CKD stage: Kidney Disease Outcomes Quality Initiative (KDOQI) CKD stages 3, 4, or 5 defined by electronic eGFR using the CKD Epidemiology Collaboration (CKD-EPI) formula.
* Erythropoietin-stimulating agents (ESAs)/Hgb: Group 1 (not using ESAs): No ESA use within the 6 weeks prior to screening and no ESA use between screening and randomization (Day 1). Group 2 (ESA users): Use of any approved ESA for the 6 weeks prior to screening and continuing between screening and randomization.
* For Group 1 (not using ESAs), Hgb concentration at Week -8 and Week 1 should be 8 to 10 gram per deciliter (g/dL). For Group 2 (ESA users), Hgb concentration at Week -8 should be 8 to 12 g/dL and at Week 1 should be 8 to 11 g/dL.
* >=80% and <=120% compliance with placebo during run-in period.
* Informed consent (screening only): capable of giving signed informed consent which includes compliance with the requirements and restrictions.

Exclusion Criteria:

* Dialysis: On dialysis or clinical evidence of impending need to initiate dialysis within 90 days after study start (Day 1).
* Kidney transplant: Planned living-related or living-unrelated kidney transplant within 52 weeks after study start (Day 1).
* Ferritin: <=100 nanograms (ng)/milliliter (mL) (<=100 micrograms/liter [L]) at screening.
* Transferrin saturation (TSAT) (screening only): <=20%.
* Aplasias: History of bone marrow aplasia or pure red cell aplasia.
* Other causes of anemia: untreated pernicious anemia, thalassemia major, sickle cell disease or myelodysplastic syndrome.
* Gastrointestinal (GI) bleeding: Evidence of actively bleeding gastric, duodenal, or esophageal ulcer disease or clinically significant GI bleeding <=4 weeks prior to screening through to randomization (Day 1).
* MI or acute coronary syndrome: <=4 weeks prior to screening through to randomization (Day 1).
* Stroke or transient ischemic attack: <=4 weeks prior to screening through to randomization (Day 1).
* Heart failure (HF): Chronic Class IV HF, as defined by the New York Heart Association (NYHA) functional classification system.
* Current uncontrolled hypertension: Current uncontrolled hypertension as determined by the investigator.
* Bazett's corrected QT interval (QTcB) (Day 1): QTcB >500 millisecond (msec), or QTcB >530 msec in subjects with bundle branch block. There is no Q-T Interval Corrected for Heart Rate (QTc) exclusion for subjects with a predominantly ventricular paced rhythm.
* Alanine transaminase (ALT): >2x upper limit of normal (ULN) at screening.
* Bilirubin: >1.5xULN at screening.
* Current unstable liver or biliary disease per investigator assessment, generally defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices, persistent jaundice, or cirrhosis.
* Malignancy: History of malignancy within the 2 years prior to screening through to randomization (Day 1) or currently receiving treatment for cancer, or complex kidney cyst (example [e.g.] Bosniak Category II F, III or IV) > 3 centimeter (cm); with the exception of localized squamous cell or basal cell carcinoma of the skin that has been definitively treated >=4 weeks prior to screening.
* Severe allergic reactions: History of severe allergic or anaphylactic reactions or hypersensitivity to excipients in the investigational product, or darbepoetin alfa.
* Drugs and supplements: Use of strong inhibitors of Cytochrome P4502C8 (CYP2C8) (e.g., gemfibrozil) or strong inducers of CYP2C8 (e.g., rifampin/rifampicin).
* Other study participation: Use of other investigational agent or device prior to screening through to randomization (Day 1). At screening, this exclusion applies to use of the investigational agent within 30 days or within five half lives (whichever is longer).
* Prior treatment with daprodustat: Any prior treatment with daprodustat for treatment duration of >30 days.
* Females only: Subject is pregnant [as confirmed by a positive urine human chorionic gonadotrophin (hCG) test for females of reproductive potential (FRP) only], subject is breastfeeding, or subject is of reproductive potential and does not agree to follow one of the contraceptive options.
* Other Conditions: Any other condition, clinical or laboratory abnormality, or examination finding that the investigator considers would put the subject at unacceptable risk, which may affect study compliance (e.g., intolerance to darbepoetin alfa) or prevent understanding of the aims or investigational procedures or possible consequences of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3872 (Actual)
Dates: Start 2016-09-27 (Actual); Primary Completion 2021-04-19 (Actual); Study Completion 2021-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (470):
- United States (131):
  - GSK Investigational Site, Andalusia, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Azusa, California
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Chula Vista, California
  - GSK Investigational Site, Cudahy, California
  - GSK Investigational Site, El Centro, California
  - GSK Investigational Site, Escondido, California
  - GSK Investigational Site, Glendale, California
  - GSK Investigational Site, Granada Hills, California
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, La Palma, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Montebello, California
  - GSK Investigational Site, National City, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Luis Obispo, California
  - GSK Investigational Site, Simi Valley, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Whittier, California
  - GSK Investigational Site, Middlebury, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Cutler Bay, Florida
  - GSK Investigational Site, Doral, Florida
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Homestead, Florida
  - GSK Investigational Site, Hudson, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Lauderdale Lakes, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Miami Gardens, Florida
  - GSK Investigational Site, Miami Lakes, Florida
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Port Charlotte, Florida
  - GSK Investigational Site, South Miami, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Temple Terrace, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Crystal Lake, Illinois
  - GSK Investigational Site, Mount Prospect, Illinois
  - GSK Investigational Site, Quincy, Illinois
  - GSK Investigational Site, Springfield, Illinois
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Jeffersonville, Indiana
  - GSK Investigational Site, Michigan City, Indiana
  - GSK Investigational Site, Des Moines, Iowa
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Hutchinson, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Baton Rouge, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Potomac, Maryland
  - GSK Investigational Site, Takoma Park, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, Kalamazoo, Michigan
  - GSK Investigational Site, Pontiac, Michigan
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Tupelo, Mississippi
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, North Platte, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Flushing, New York
  - GSK Investigational Site, Laurelton, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Ridgewood, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Yonkers, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Rocky Mount, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Grand Forks, North Dakota
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Mentor, Ohio
  - GSK Investigational Site, Lawton, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Roseburg, Oregon
  - GSK Investigational Site, Bethlehem, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Cordova, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Corsicana, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lufkin, Texas
  - GSK Investigational Site, McAllen, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Waxahachie, Texas
  - GSK Investigational Site, Alexandria, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Salem, Virginia
  - GSK Investigational Site, Bluefield, West Virginia
- Argentina (13):
  - GSK Investigational Site, Ciudad Evita, Buenos Aires
  - GSK Investigational Site, Coronel Suárez, Buenos Aires
  - GSK Investigational Site, Junín, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
  - GSK Investigational Site, Pergamino, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Corrientes
  - GSK Investigational Site, Formosa
  - GSK Investigational Site, La Plata
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, Morón
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (14):
  - GSK Investigational Site, Garran, Australian Capital Territory
  - GSK Investigational Site, Concord, New South Wales
  - GSK Investigational Site, Gosford, New South Wales
  - GSK Investigational Site, Kingswood, New South Wales
  - GSK Investigational Site, Kogarah, New South Wales
  - GSK Investigational Site, Randwick, New South Wales
  - GSK Investigational Site, St Leonards, New South Wales
  - GSK Investigational Site, Wollongong, New South Wales
  - GSK Investigational Site, Nambour, Queensland
  - GSK Investigational Site, Melbourne, Victoria
  - GSK Investigational Site, Reservoir, Victoria
  - GSK Investigational Site, St Albans, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
  - GSK Investigational Site, Liverpool
- Belgium (10):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Baudour
  - GSK Investigational Site, Bruges
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Ieper
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Roeselare
  - GSK Investigational Site, Ronse
  - GSK Investigational Site, Sint-Niklaas
- Brazil (12):
  - GSK Investigational Site, Salvador, Estado de Bahia
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Passo Fundo, Rio Grande do Sul
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São José do Rio Preto, São Paulo
  - GSK Investigational Site, Votuporanga, São Paulo
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Brasília
  - GSK Investigational Site, Feira de Santana
  - GSK Investigational Site, Joinville
  - GSK Investigational Site, Juiz de Fora
  - GSK Investigational Site, São Paulo
- Bulgaria (13):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Burgas
  - GSK Investigational Site, Dobrich
  - GSK Investigational Site, Gabrovo
  - GSK Investigational Site, Lom
  - GSK Investigational Site, Pazardzhik
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sliven
  - GSK Investigational Site, Smolyan
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Varna
  - GSK Investigational Site, Veliko Tarnovo
- Canada (9):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Greenfield Park, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Colombia (5):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Cali
  - GSK Investigational Site, Floridablanca
  - GSK Investigational Site, Medellín
- Czechia (9):
  - GSK Investigational Site, Beroun
  - GSK Investigational Site, Český Krumlov
  - GSK Investigational Site, Ivančice
  - GSK Investigational Site, Jilemnice
  - GSK Investigational Site, Mariánské Lázně
  - GSK Investigational Site, Nový Jičín
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Sokolov
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Holstebro
  - GSK Investigational Site, Kolding
  - GSK Investigational Site, Odense C
- Estonia (3):
  - GSK Investigational Site, Jämejala Village
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (9):
  - GSK Investigational Site, Annonay
  - GSK Investigational Site, Boulogne-Billancourt
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Mulhouse
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Saint-Ouen
- Germany (9):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Cloppenburg, Lower Saxony
  - GSK Investigational Site, Düsseldorf, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Kaiserslautern, Rhineland-Palatinate
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Cologne
  - GSK Investigational Site, Wiesbaden
- Greece (11):
  - GSK Investigational Site, Alexandroupoli
  - GSK Investigational Site, Arta
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Efkarpia
  - GSK Investigational Site, Heraklion-Crete
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Komotini
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Melíssia
  - GSK Investigational Site, Pátrai
  - GSK Investigational Site, Thessaloniki
- Hong Kong (4):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Lai Chi Kok
  - GSK Investigational Site, New Territories
  - GSK Investigational Site, Tsuen Wan
- Hungary (8):
  - GSK Investigational Site, Baja
  - GSK Investigational Site, Balatonfüred
  - GSK Investigational Site, Esztergom
  - GSK Investigational Site, Kecskemét
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Salgótarján
  - GSK Investigational Site, Szigetvár
- India (20):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Calicut
  - GSK Investigational Site, Chandigarh
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Chennai, Tamil Nadu
  - GSK Investigational Site, Delhi
  - GSK Investigational Site, Ghaziabad
  - GSK Investigational Site, Gūrgaon
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, Manipal
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nadiād
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Secunderabad
  - GSK Investigational Site, Trivandrum
- Israel (8):
  - GSK Investigational Site, Ashkelon
  - GSK Investigational Site, Hadera
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Nahariya
  - GSK Investigational Site, Nazareth
  - GSK Investigational Site, Poria – Neve Oved
  - GSK Investigational Site, Ẕerifin
- Italy (13):
  - GSK Investigational Site, Foggia, Apulia
  - GSK Investigational Site, Catanzaro, Calabria
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Piacenza, Emilia-Romagna
  - GSK Investigational Site, Reggio Emilia, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Lecco, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Cagliari, Sardinia
  - GSK Investigational Site, Imola
  - GSK Investigational Site, Mestre
- Malaysia (7):
  - GSK Investigational Site, Alor Star
  - GSK Investigational Site, George Town
  - GSK Investigational Site, Ipoh
  - GSK Investigational Site, Kuala Lumpur
  - GSK Investigational Site, Kuala Pahang
  - GSK Investigational Site, Kuantan
  - GSK Investigational Site, Lumut
- Mexico (19):
  - GSK Investigational Site, Saltillo, Coahuila
  - GSK Investigational Site, Torreón, Coahuila
  - GSK Investigational Site, Durango, Durango
  - GSK Investigational Site, León, Guanajuato
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Cuernavaca, Morelos
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Querétaro City, Querétaro
  - GSK Investigational Site, Culiacán, Sinaloa
  - GSK Investigational Site, Mazatlán, Sinaloa
  - GSK Investigational Site, Ciudad de Mexico, State of Mexico
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, Aguascalientes
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Culiacán
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Tlalnepantla
  - GSK Investigational Site, Veracruz
  - GSK Investigational Site, Zapopan, Jalisco
- Netherlands (3):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Deventer
  - GSK Investigational Site, Rotterdam
- New Zealand (5):
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Hastings
  - GSK Investigational Site, Otahuhu
  - GSK Investigational Site, Takapuna, Auckland
- Philippines (9):
  - GSK Investigational Site, Baguio City, Benguet
  - GSK Investigational Site, Cebu City
  - GSK Investigational Site, Dasmariñas
  - GSK Investigational Site, Iloilo City
  - GSK Investigational Site, Manila
  - GSK Investigational Site, Pasig
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, San Juan City
  - GSK Investigational Site, Sto Tomas
- Poland (10):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Brzeg
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Kielce
  - GSK Investigational Site, Kołobrzeg
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Radom
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Żyrardów
- Portugal (5):
  - GSK Investigational Site, Amadora
  - GSK Investigational Site, Aveiro
  - GSK Investigational Site, Covilha
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Torres Novas
- Romania (4):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Timișoara
- Russia (13):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Mytischi
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Podolsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Volzhsky
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Singapore, Singapore
- South Africa (3):
  - GSK Investigational Site, Port Elizabeth, Eastern Cape
  - GSK Investigational Site, Cape Town
  - GSK Investigational Site, Somerset West
- South Korea (14):
  - GSK Investigational Site, Anyang-Si, Gyeonggi-do
  - GSK Investigational Site, Bucheon-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Goyang-si
  - GSK Investigational Site, Ilsanseo-gu, Goyang-si,
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Seongnam
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
  - GSK Investigational Site, Uijeongbu-si
  - GSK Investigational Site, Wŏnju
- Spain (12):
  - GSK Investigational Site, Majadahonda, Madrid
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Burela de Cabo
  - GSK Investigational Site, Cáceres
  - GSK Investigational Site, Ciudad Real
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Mollet del Vallès
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
- Sweden (3):
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Taiwan (6):
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Keelung
  - GSK Investigational Site, New Taipei City
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan Hsien
- Thailand (5):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Bangkoknoi
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Pathum Thani
- Turkey (Türkiye) (7):
  - GSK Investigational Site, Adana
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Antalya
  - GSK Investigational Site, Edirne
  - GSK Investigational Site, Eskişehir
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Kayseri
- Ukraine (14):
  - GSK Investigational Site, Cherkasy
  - GSK Investigational Site, Chernihiv
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Ivano-Frankivsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kherson
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Lutsk
  - GSK Investigational Site, Mykolaiv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Ternopil
  - GSK Investigational Site, Zaporizhzhia
  - GSK Investigational Site, Zhytomyr
- United Kingdom (21):
  - GSK Investigational Site, Stevenage, Hertfordshire
  - GSK Investigational Site, Preston, Lancashire
  - GSK Investigational Site, Hampstead, London
  - GSK Investigational Site, Liverpool, Merseyside
  - GSK Investigational Site, Wolverhampton, West Midlands
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Cardiff
  - GSK Investigational Site, Derby
  - GSK Investigational Site, Doncaster
  - GSK Investigational Site, Fife
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Hull
  - GSK Investigational Site, Leeds
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Oxford
  - GSK Investigational Site, Salford
  - GSK Investigational Site, York
- Vietnam (4):
  - GSK Investigational Site, Haiphong
  - GSK Investigational Site, Hanoi
  - GSK Investigational Site, Hà Nội
  - GSK Investigational Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD is made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency

REFERENCES:
- [Background] Ajay K. Singh, Kevin Carroll, John J. V. McMurray, Scott Solomon, Vivekanand Jha, Kirsten L. Johansen, Renato D. Lopes, Iain C. Macdougall, Gregorio T. Obrador, Sushrut S. Waikar, Christoph Wanner, David C. Wheeler, Andrzej Wiecek, Allison Blackorby, Borut Cizman, Alexander R. Cobitz, Rich Davies, Tara L. DiMino, Lata Kler, Amy M. Meadowcroft, Lin Taft, Vlado Perkovic for the ASCEND-ND Study Group. DAPRODUSTAT FOR THE TREATMENT OF ANEMIA IN PATIENTS NOT UNDERGOING DIALYSIS. N Engl J Med. 2021; DOI: 10.1056/NEJMoa2113380 PMID: 34739196
- [Background] Perkovic V, Blackorby A, Cizman B, Carroll K, Cobitz AR, Davies R, DiMino TL, Jha V, Johansen KL, Lopes RD, Kler L, Macdougall IC, McMurray JJV, Meadowcroft AM, Obrador GT, Solomon S, Taft L, Wanner C, Waikar SS, Wheeler DC, Wiecek A, Singh AK. The ASCEND-ND trial: study design and participant characteristics. Nephrol Dial Transplant. 2022 Oct 19;37(11):2157-2170. doi: 10.1093/ndt/gfab318. PMID 34865143
- [Derived] Cunningham JW, Claggett BL, Lopes RD, McMurray JJV, Perkovic V, Carroll K, Hiemstra T, Khavandi K, Lukas MA, Ranganathan P, Shannon J, van Adelsberg J, Singh AK, Solomon SD. Daprodustat and Heart Failure in CKD. J Am Soc Nephrol. 2024 May 1;35(5):607-617. doi: 10.1681/ASN.0000000000000321. Epub 2024 Feb 22. PMID 38383961
- [Derived] Singh AK, McCausland FR, Claggett BL, Wanner C, Wiecek A, Atkins MB, Carroll K, Perkovic V, McMurray JJV, Wittes J, Snapinn S, Blackorby A, Meadowcroft A, Barker T, DiMino T, Mallett S, Cobitz AR, Solomon SD. Analysis of on-treatment cancer safety events with daprodustat versus conventional erythropoiesis-stimulating agents-post hoc analyses of the ASCEND-ND and ASCEND-D trials. Nephrol Dial Transplant. 2023 Jul 31;38(8):1890-1897. doi: 10.1093/ndt/gfac342. PMID 36565721
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Singh AK, Carroll K, McMurray JJV, Solomon S, Jha V, Johansen KL, Lopes RD, Macdougall IC, Obrador GT, Waikar SS, Wanner C, Wheeler DC, Wiecek A, Blackorby A, Cizman B, Cobitz AR, Davies R, DiMino TL, Kler L, Meadowcroft AM, Taft L, Perkovic V; ASCEND-ND Study Group. Daprodustat for the Treatment of Anemia in Patients Not Undergoing Dialysis. N Engl J Med. 2021 Dec 16;385(25):2313-2324. doi: 10.1056/NEJMoa2113380. Epub 2021 Nov 5. PMID 34739196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted across 39 countries. Participants were randomized to receive either daprodustat or darbepoetin alfa.
Pre-assignment Details: A total of 3872 participants were enrolled in the study.
Groups:
- Daprodustat: Participants received placebo tablets orally once daily in run-in period from Week-4 up to randomization (Day 1) and subsequently received treatment with daprodustat film-coated tablets at dose levels ranging from 1, 2, 4, 6, 8, 10, 12, 16 and 24 milligrams (mg) orally once daily up to 51.1 month. Study treatment was dose-titrated to achieve and maintain hemoglobin (Hgb) in the target range (10 to 11 grams per deciliter [g/dL]).
- Darbepoetin Alfa: Participants received placebo tablets orally once daily in run-in period from Week-4 up to randomization (Day 1) and subsequently received treatment with darbepoetin alfa as prefilled syringes (PFS) for subcutaneous or intravenous (IV) injection at 4-weekly total dose levels ranging from 20, 30, 40, 60, 80, 100, 150, 200, 300 and 400 microgram (mcg) up to 51.1 month. Darbepoetin alfa IV injection was administered to participants undergoing hemodialysis. Study treatment was dose-titrated to achieve and maintain Hgb in the target range (10 to 11 g/dL).
Period: Run-in Period: Placebo (Week-4 to Day 1)
Arm/Group | Daprodustat | Darbepoetin Alfa
Started | 1937 | 1935
Completed | 1937 | 1935
Not Completed | 0 | 0
Period: Treatment Period (51.1 Month)
Arm/Group | Daprodustat | Darbepoetin Alfa
Started | 1937 | 1935
Completed | 1873 | 1870
Not Completed | 64 | 65
Not completed — Other | 1 | 0
Not completed — Investigator Site Closed | 6 | 13
Not completed — Withdrawal by Subject | 32 | 23
Not completed — Lost to Follow-up | 25 | 29

BASELINE CHARACTERISTICS:
Population: All Randomized (Intent-to-treat [ITT]) Population comprised of all randomized participants. Participants were analyzed according to the treatment to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Daprodustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 1937 | 1935 | 3872
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.8 (14.03) | 64.9 (13.83) | 64.8 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1102 | 1071 | 2173
  Male | 835 | 864 | 1699
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 88 | 100 | 188
  Asian - Central/South Asian Heritage | 58 | 71 | 129
  Asian - East Asian Heritage | 245 | 232 | 477
  Asian - Japanese Heritage | 5 | 3 | 8
  Asian - South East Asian Heritage | 216 | 229 | 445
  Black or African American | 183 | 185 | 368
  Native Hawaiian or Other Pacific Islander | 7 | 7 | 14
  White - Arabic/North African Heritage | 19 | 18 | 37
  White - White/Caucasian/European Heritage | 1079 | 1037 | 2116
  Mixed Asian Race | 1 | 2 | 3
  Mixed Race | 36 | 51 | 87

OUTCOME MEASURES:

1. Primary Outcome: Time to First Occurrence of Adjudicated Major Adverse Cardiovascular Event (MACE) During Cardiovascular (CV) Events Follow-up Time Period (Non-inferiority Analysis)
Description: Time to MACE defined as time to first occurrence of Clinical Events Committee (CEC) adjudicated MACE (composite of all-cause mortality, non-fatal myocardial infarction [MI] and non-fatal stroke) was analyzed using a Cox proportional hazards regression model with treatment group, current erythropoiesis-stimulating agents (ESA) use at randomization and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) plus (+) 1. The incidence rate per 100 person years calculated as (100 multiplied [*] number of participants with at least 1 event) divided by [/] first event person-years) is presented along with 95 percent (%) confidence interval (CI). First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 10.86 [9.80 to 12.02] | 10.63 [9.58 to 11.77]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — Non-inferiority was achieved if the upper limit of the two-sided 95% CI for the hazard ratio was below the pre-specified non-inferiority margin of 1.25; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.89 to 1.19] — Hazard ratio was estimated using a Cox proportional hazard regression model with treatment group, current ESA use at randomization, and region as covariates

2. Primary Outcome: Mean Change From Baseline in Hgb Levels Over the Evaluation Period (Week 28 to Week 52)
Description: Blood samples were collected from participants for Hgb measurements. Hgb during the evaluation period was defined as the mean of all available post-randomization Hgb values (on and off-treatment) during the evaluation period (Week 28 to Week 52). For the primary analysis missing post-Baseline Hgb values were imputed using pre-specified multiple imputation methods. Change from Baseline was defined as post-Baseline value minus (-) Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. Analysis was performed using the Analysis of covariance (ANCOVA) model with terms for treatment, Baseline Hgb, current ESA use and region.
Time Frame: Baseline (Pre-dose on Day 1) and evaluation period (Week 28 to Week 52)
Population: All Randomized (ITT) Population.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Grams per deciliter | 0.74 (0.019) | 0.66 (0.019)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% CI for the treatment difference was greater than -0.75 g/dL; Least square (LS) mean difference = 0.08, 95% CI 2-sided [0.03 to 0.13]

3. Secondary Outcome: Time to First Occurrence of Adjudicated MACE During CV Events Follow-up Time Period (Superiority Analysis)
Description: Time to MACE defined as the time to first occurrence of CEC adjudicated MACE was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariate. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period. This endpoint was adjusted for multiplicity using the Holm-Bonferonni method.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 10.86 [9.80 to 12.02] | 10.63 [9.58 to 11.77]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.670884, Wald test — The p-value was compared against 0.008333 based on the Holm-Bonferonni adjustment; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.89 to 1.19] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Time to First Occurrence of Adjudicated MACE or Thromboembolic Event During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MACE or thromboembolic event (vascular access thrombosis, symptomatic deep vein thrombosis or symptomatic pulmonary embolism) was analyzed using a Cox proportional hazards regression model with with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period. This endpoint was adjusted for multiplicity using the Holm-Bonferonni method.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 12.34 [11.19 to 13.57] | 11.77 [10.65 to 12.98]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.800813, Wald test — The p-value was compared against 0.012500 based on the Holm-Bonferonni adjustment; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.93 to 1.22] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Time to First Occurrence of Adjudicated MACE or Hospitalization for Heart Failure During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MACE or hospitalization for heart failure was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period. This endpoint was adjusted for multiplicity using the Holm-Bonferonni method.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 13.16 [11.97 to 14.44] | 12.22 [11.08 to 13.46]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.886195, Wald test — The p-value was compared against 0.025000 based on the Holm-Bonferonni adjustment; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.95 to 1.24] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Time to First Occurrence of Chronic Kidney Disease (CKD) Progression During CV Events Follow-up Time Period
Description: Progression of CKD defined as: 40% decline in estimated glomerular filtration rate (eGFR) from Baseline or end stage renal disease (ESRD) as defined by either initiating chronic dialysis for >=90 days or not initiating chronic dialysis when dialysis is indicated or kidney transplantation. Time to first occurrence of CKD progression was analyzed using Fine and Gray's proportional subdistribution hazard regression model with treatment group, Baseline ESA use and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) +1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed. Additionally, this analysis population was restricted to those with a Baseline eGFR >=15milliliter per minute (mL/min).
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1220 | 1265
Events per 100 person years | 17.55 [15.74 to 19.51] | 17.76 [15.97 to 19.70]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.369470, Wald test; Subdistribution hazard ratio = 0.98, 95% CI 2-sided [0.84 to 1.13] — Subdistribution hazard ratio was estimated using Fine and Gray's proportional subdistribution hazard regression model with treatment group, Baseline ESA use, and region as covariates

7. Secondary Outcome: Time to First Occurrence of Adjudicated All-Cause Mortality During Vital Status for Follow-up Time Period
Description: Time to first occurrence of adjudicated all-cause mortality was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the vital status follow-up time period.
Time Frame: Up to 4.3 person-years for vital status follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 8.35 [7.43 to 9.35] | 8.27 [7.35 to 9.26]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6197, Wald test; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.87 to 1.20] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Time to First Occurrence of Adjudicated CV Mortality During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated CV mortality was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 3.02 [2.48 to 3.65] | 2.55 [2.06 to 3.13]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8976, Wald test; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.91 to 1.58] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Time to First Occurrence of Adjudicated Myocardial Infarction (MI) (Fatal and Non-Fatal) During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MI (fatal and non-fatal) was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 2.94 [2.40 to 3.56] | 2.76 [2.24 to 3.36]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6581, Wald test; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.80 to 1.40] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Time to First Occurrence of Adjudicated Stroke (Fatal and Non-Fatal) During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated stroke (fatal and non-fatal) was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 1.26 [0.92 to 1.69] | 0.95 [0.66 to 1.33]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8940, Wald test; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [0.85 to 2.07] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Number of Participants With Adjudicated MACE or Hospitalization for Heart Failure (Recurrent Events Analysis)
Description: Number of participants with adjudicated MACE or hospitalization for heart failure (recurrent events analysis) is presented, categorized by number of occurrences of adjudicated MACE or hospitalization for heart failure per participant.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Participants
  Occurrences per participant: 0 | 1493 | 1518
  Occurrences per participant: 1 | 318 | 317
  Occurrences per participant: 2 | 76 | 64
  Occurrences per participant: 3 | 26 | 22
  Occurrences per participant: 4 | 14 | 9
  Occurrences per participant: 5 | 5 | 3
  Occurrences per participant: 6 | 1 | 0
  Occurrences per participant: 7 | 4 | 1
  Occurrences per participant: 8 | 0 | 1
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9422, Chi-squared; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.98 to 1.23] — Overall HR is presented using Model 1. Model 1 assumed a common treatment effect, regardless of number of events experienced. HR was estimated using a Prentice, Williams and Peterson(PWP) model, with treatment, dialysis type and region as covariates
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8862, Chi-squared; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.95 to 1.24] — First Event Hazard ratio is presented using Model 2. Model 2 assumed treatment effect differs by number of events experienced. Hazard Ratio (HR) was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6789, Chi-squared; Hazard Ratio (HR) = 1.07, 95% CI 2-sided [0.82 to 1.39] — Second Event Hazard ratio is presented using Model 2. Model 2 assumed treatment effect differs by number of events experienced. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9016, Chi-squared; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.85 to 2.19] — Third Event Hazard ratio is presented using Model 2. Model 2 assumed treatment effect differs by number of events experienced. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 5: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8862, Chi-squared; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.95 to 1.24] — First Event Hazard ratio is presented using Model 3. Model 3 assumed treatment effect for first event differs from a common effect for subsequent events. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates
Statistical Analysis 6: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8989, Chi-squared; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.92 to 1.46] — Subsequent Event Hazard ratio is presented using Model 3. Model 3 assumed treatment effect for first event differs from a common effect for subsequent events. HR was estimated using a PWP model, with treatment, dialysis type and region as covariates

12. Secondary Outcome: Time to First Occurrence of Adjudicated CV Mortality or Non-Fatal MI During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated CV mortality or non-fatal MI was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 5.36 [4.62 to 6.18] | 4.98 [4.27 to 5.77]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7673, Wald test; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.88 to 1.33] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Time to First Occurrence of All-Cause Hospitalization During CV Events Follow-up Time Period
Description: All-cause hospitalization events were hospital admissions recorded on the hospitalization electronic case report form (eCRF) form with a hospitalization duration >=24 hours. Time to first occurrence of all-cause hospitalization was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 41.13 [38.59 to 43.80] | 38.99 [36.54 to 41.56]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8601, Wald test; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.96 to 1.15] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Time to First Occurrence of All-Cause Hospital Re-admission Within 30 Days During CV Events Follow-up Time Period
Description: All-cause hospital re-admissions within 30days are defined as hospital admissions recorded on hospitalization electronic case record form with hospitalization duration of >=24 hours and admission date within 30days following previous discharge date of all-cause hospitalization event, where previous hospitalization was >=24hours.Time to first occurrence of all-cause hospital re-admission within 30days was analyzed using Cox proportional hazards regression model with treatment group, current ESA use at randomization and region as covariates.Time to the first occurrence was computed as(event date - randomization date)+1. Incidence rate per 100 person years calculated as(100*number of participants with at least 1event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event+cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 7.78 [6.87 to 8.79] | 7.55 [6.65 to 8.55]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6207, Wald test; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.86 to 1.22] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Time to First Occurrence of Adjudicated MACE or Hospitalization for Heart Failure or Thromboembolic Events During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated MACE or hospitalization for heart failure or thromboembolic events were analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 14.60 [13.33 to 15.96] | 13.32 [12.11 to 14.61]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9393, Wald test; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.97 to 1.26] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Time to First Occurrence of Adjudicated Hospitalization for Heart Failure During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated hospitalization for heart failure was analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 4.05 [3.41 to 4.78] | 3.30 [2.73 to 3.96]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9412, Wald test; Hazard Ratio (HR) = 1.22, 95% CI 2-sided [0.95 to 1.56] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Time to First Occurrence of Adjudicated Thromboembolic Events During CV Events Follow-up Time Period
Description: Time to first occurrence of adjudicated thromboembolic events were analyzed using a Cox proportional hazards regression model with treatment group, current ESA use at randomization, and region as covariates. Time to the first occurrence was computed as (event date minus randomization date) + 1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Events per 100 person years | 1.81 [1.39 to 2.31] | 1.43 [1.07 to 1.89]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8994, Wald test; Hazard Ratio (HR) = 1.27, 95% CI 2-sided [0.88 to 1.84] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Time to First Occurrence of Confirmed 40% Decline in eGFR During CV Events Follow-up Time Period
Description: Time to first occurrence of confirmed 40% decline in eGFR was analyzed using a Fine & Gray's proportional subdistribution hazard regression model with treatment group, Baseline ESA use and region as covariates. Time to the first occurrence was computed as (event date minus randomization date)+1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1220 | 1265
Events per 100 person years | 8.21 [7.04 to 9.52] | 8.90 [7.69 to 10.24]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.2073, Wald test; Subdistribution hazard ratio = 0.92, 95% CI 2-sided [0.75 to 1.13] — Subdistribution hazard ratio was estimated using Fine & Gray's proportional subdistribution hazard regression model with treatment group, Baseline ESA use, and region as covariates

19. Secondary Outcome: Time to First Occurrence of Chronic Dialysis During CV Events Follow-up Time Period
Description: Time to first occurrence of chronic dialysis was analyzed using a Fine & Gray's proportional subdistribution hazard regression model with treatment group, Baseline ESA use and region as covariates. Chronic dialysis is defined by either initiating dialysis for >=90 days or not initiating chronic dialysis when dialysis is indicated. Time to the first occurrence was computed as (event date minus randomization date)+1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1220 | 1265
Events per 100 person years | 12.20 [10.74 to 13.81] | 12.06 [10.63 to 13.62]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5068, Wald test; Subdistribution hazard ratio = 1.00, 95% CI 2-sided [0.84 to 1.19] — [estimate comment as in outcome 18, analysis 1]

20. Secondary Outcome: Time to First Occurrence of Kidney Transplant During CV Events Follow-up Time Period
Description: Time to first occurrence of kidney transplant were analyzed using a Fine & Gray's proportional subdistribution hazard regression model with treatment group, Baseline ESA use and region as covariates. Time to the first occurrence was computed as (event date minus randomization date)+1. The incidence rate per 100 person years calculated as (100*number of participants with at least 1 event)/first event person-years) is presented along with 95% CI. First event person years=(cumulative total time to first event for participants who have the event + cumulative total of censored time for participants without the event)/365.25, based on the CV follow-up time period.
Time Frame: Up to 4.3 person-years for CV follow-up time period
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Events per 100 person years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1220 | 1265
Events per 100 person years | 1.00 [0.63 to 1.50] | 1.14 [0.75 to 1.66]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3285, Wald test; Subdistribution hazard ratio = 0.88, 95% CI 2-sided [0.51 to 1.54] — [estimate comment as in outcome 18, analysis 1]

21. Secondary Outcome: Change From Baseline in Post-randomization Hgb Levels at Week 52
Description: Blood samples were collected from participants for Hgb measurements. Change from Baseline was defined as post-randomization value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. Analysis was performed using mixed model repeated measures (MMRM) model fitted from Baseline up to Week 52, excluding values collected during the stabilization period, with factors for treatment, time, current ESA use, region, Baseline Hgb and Baseline Hgb by time and treatment by time interactions.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Grams per deciliter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1557 | 1556
Grams per deciliter | 0.76 (0.029) | 0.73 (0.029)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% CI for the treatment difference was greater than the pre-specified non-inferiority margin of -0.75 g/dL; LS mean difference = 0.03, 95% CI 2-sided [-0.05 to 0.11]

22. Secondary Outcome: Number of Hgb Responders in the Hgb Analysis Range (10 to 11.5 Grams/Deciliter) During Evaluation Period (Week 28 to Week 52)
Description: Mean Hgb during the evaluation period was defined as the mean of all evaluable Hgb values during the evaluation period (Week 28 to Week 52) including any evaluable unscheduled Hgb values that were taken during this time period. Hgb responders were defined as participants with a mean Hgb during the evaluation period that falls within the Hgb analysis range of 10-11.5 g/dL.
Time Frame: Week 28 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1491 | 1520
Participants | 1167 | 1063
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in response rate = 8.3, 95% CI 2-sided [5.2 to 11.4] — Cochran-Mantel-Haenszel (CMH) test adjusted for current ESA use and region was used to compare the number of responders between the treatment groups

23. Secondary Outcome: Percentage of Time With Hgb in the Analysis Range (10 to 11.5 Grams/Deciliter) During Evaluation Period (Week 28 to Week 52): Non-inferiority Analysis
Description: Percentage of days for which a participant's Hgb was within the analysis range of 10-11.5 g/dL (both inclusive) during the evaluation period (Week 28 to Week 52), including any unscheduled evaluable Hgb values that were taken during this time period was calculated. Percentage of time in the analysis range during evaluation period is calculated as time in range during the evaluation period / [Earlier of (Date of the last evaluable Hgb value, Week 52 visit date) - Later of (Date of the first evaluable Hgb value that between Week 16 and Week 52 inclusive, Week 28 visit date)].
Time Frame: Week 28 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1461 | 1483
Percentage of days | 70.5 [0.0 to 100.0] | 63.2 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — Non-inferiority was to be established if the lower limit of the two-sided 95% confidence interval for the treatment difference was greater than non-inferiority margin of -15%; Mean Difference (Final Values) = 4.57, 95% CI 2-sided [2.04 to 7.11] — Hodges-Lehmann estimate of the treatment difference (daprodustat-darbepoetin alfa) and associated two-sided asymptotic 95% CI is presented

24. Secondary Outcome: Percentage of Time With Hgb in the Analysis Range (10 to 11.5 Grams/Deciliter) During Evaluation Period (Week 28 to Week 52): Superiority Analysis
Description: as for outcome 23
Time Frame: Week 28 to Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1461 | 1483
Percentage of days | 70.5 [0.0 to 100.0] | 63.2 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p < 0.0001, van Elteren test; Probability = 0.55, 95% CI 2-sided [0.53 to 0.57] — Mann-Whitney estimate (Probability) of the treatment effect has been presented

25. Secondary Outcome: Percentage of Time With Hgb in the Analysis Range (10 to 11.5 Grams/Deciliter) During Maintenance Period (Week 28 to End of Study): Non-inferiority Analysis
Description: Percentage of days for which a participant's Hgb was within the analysis range of 10-11.5 g/dL (both inclusive) during the maintenance period (Week 28 to end of study), including any unscheduled evaluable Hgb values that were taken during this time period was calculated. Percentage of time in the analysis range during maintenance period is calculated as time in range during the maintenance period / [Earlier of (Date of the last evaluable Hgb value, End of study date)- Later of (Date of the first evaluable Hgb value that is on or after week 16, Week 28 visit date)].
Time Frame: Week 28 to end of study (4.3 person-years for follow-up time period)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1469 | 1489
Percentage of days | 66.1 [0.0 to 100.0] | 62.1 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Non-Inferiority — [test comment as in outcome 23, analysis 1]; Median Difference (Final Values) = 3.94, 95% CI 2-sided [1.90 to 5.91] — [estimate comment as in outcome 23, analysis 1]

26. Secondary Outcome: Percentage of Time With Hemoglobin in the Analysis Range (10 to 11.5 Grams/Deciliter) During Maintenance Period (Week 28 to End of Study): Superiority Analysis
Description: as for outcome 25
Time Frame: Week 28 to end of study (4.3 person-years for follow-up time period)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Median (Full Range); unit: Percentage of days
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1469 | 1489
Percentage of days | 66.1 [0.0 to 100.0] | 62.1 [0.0 to 100.0]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p < 0.0001, van Elteren test; Probability = 0.54, 95% CI 2-sided [0.52 to 0.56] — Mann-Whitney estimate (Probability) of the treatment effect has been presented

27. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP), Diastolic Blood Pressure (DBP) and Mean Arterial Blood Pressure (MAP) at Week 52
Description: SBP, DBP and MAP were measured in a seated position after at least a 5-minutes of rest. MAP is the average (BP) in an individual's arteries during a single cardiac cycle. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. Analysis was performed using MMRM model with treatment group + time + current ESA use at randomization + region + Baseline value + Baseline value*time + treatment group*time, using an unstructured covariance matrix. Data for post-dialysis BP measurements have been presented.
Time Frame: Baseline (Week -4) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1913 | 1884
Millimeter of mercury
  SBP, n=1913, 1884 | -0.62 (0.488) | -1.17 (0.479)
  DBP, n=1912, 1884: number analyzed (Participants) | 1912 | 1884
  DBP, n=1912, 1884 | 0.06 (0.267) | -0.59 (0.262)
  MAP, n=1912, 1884: number analyzed (Participants) | 1912 | 1884
  MAP, n=1912, 1884 | -0.17 (0.300) | -0.77 (0.294)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7916, MMRM; LS mean difference = 0.56, 95% CI 2-sided [-0.79 to 1.90] — The difference in change from Baseline in SBP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9581, MMRM; LS mean difference = 0.65, 95% CI 2-sided [-0.09 to 1.38] — The difference in change from Baseline in DBP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9241, MMRM; LS mean difference = 0.60, 95% CI 2-sided [-0.22 to 1.43] — The difference in change from Baseline in MAP at Week 52 was analyzed with a MMRM approach with an unstructured covariance matrix to compare the difference in LS means between arms

28. Secondary Outcome: Change From Baseline in SBP, DBP, MAP at End of Treatment
Description: SBP, DBP and MAP were measured in a seated position after at least a 5-minutes of rest. MAP is an average BP in an individual's arteries during a single cardiac cycle. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date. Analysis was performed using ANCOVA model with terms for treatment group, current ESA use at randomization, region and Baseline value. Data for post-dialysis BP measurements have been presented.
Time Frame: Baseline (Week -4) and 51.1 months
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1919 | 1884
Millimeter of mercury
  SBP, n=1919, 1884 | -1.19 (0.395) | -1.10 (0.398)
  DBP, n=1918, 1884: number analyzed (Participants) | 1918 | 1884
  DBP, n=1918, 1884 | -0.26 (0.229) | -0.38 (0.231)
  MAP, n=1918, 1884: number analyzed (Participants) | 1918 | 1884
  MAP, n=1918, 1884 | -0.57 (0.248) | -0.62 (0.251)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.4420, ANCOVA; LS mean difference = -0.08, 95% CI 2-sided [-1.18 to 1.02] — For SBP: Treatment group comparisons were based on an ANCOVA model with terms for treatment group, current ESA use at randomization, region and Baseline value
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6369, ANCOVA; LS mean difference = 0.11, 95% CI 2-sided [-0.52 to 0.75] — For DBP: Treatment group comparisons were based on an ANCOVA model with terms for treatment group, current ESA use at randomization, region and Baseline value
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5490, ANCOVA; LS mean difference = 0.04, 95% CI 2-sided [-0.65 to 0.74] — For MAP: Treatment group comparisons were based on an ANCOVA model with terms for treatment group, current ESA use at randomization, region and Baseline value

29. Secondary Outcome: Blood Pressure (BP) Exacerbation Event Rate Per 100 Participant Years
Description: BP exacerbation event (based on post-dialysis) was defined as: SBP >= 25 millimeter of mercury (mmHg) increased from Baseline or SBP >=180 mmHg; DBP >=15 mmHg increased from Baseline or DBP >=110 mmHg. The BP exacerbation events per 100 participant years was estimated using the negative binomial model with treatment, current ESA use at randomization and region as covariates and the logarithm of time on-treatment as an offset variable. Data for post-dialysis BP measurements have been presented.
Time Frame: Day 1 to end of treatment (51.1 months)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number (95% Confidence Interval); unit: Events per 100 participant years
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1919 | 1884
Events per 100 participant years | 138.50 [128.58 to 149.18] | 157.35 [146.30 to 169.23]
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.0074, Negative binomial model; Ratio of exacerbation rate = 0.88, 95% CI 2-sided [0.79 to 0.98] — Ratio of model estimated exacerbation rates and CIs estimated using negative binomial model with treatment,current ESA use at randomization and region as covariates and logarithm of time on treatment as offset variable for treatment group comparison

30. Secondary Outcome: Number of Participants With at Least One BP Exacerbation Event During Study
Description: BP exacerbation was defined as: SBP >= 25 mmHg increased from Baseline or SBP >=180 mmHg; DBP >=15 mmHg increased from Baseline or DBP >=110 mmHg. Number of participants with at least one BP exacerbation event is presented.
Time Frame: Day 1 to end of treatment (51.1 months)
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1919 | 1884
Participants | 939 | 1012

31. Secondary Outcome: Percentage of Participants Permanently Stopping Randomized Treatment Due to Meeting Rescue Criteria
Description: Percentage of participants permanently stopping randomized treatment due to meeting rescue criteria has been presented.
Time Frame: Day 1 to 51.1 months
Population: All Randomized (ITT) Population.
Measure: Number; unit: Percentage of participants
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1937 | 1935
Percentage of participants | 2.0 | 3.3
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.0113, Wald test; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.42 to 0.94] — Hazard ratio was estimated using a Cox proportional hazard regression model adjusted for treatment group, current ESA use and region

32. Secondary Outcome: Change From Baseline in On-treatment Physical Component Score (PCS) Using Short Form (SF)-36 Health-related Quality of Life (HRQoL) Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). The PCS is an average score derived from 4 domains (physical functioning, role-physical, bodily pain and general health) representing overall physical health. PCS ranges from 0 to 100; higher score represents better health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1238 | 1227
Scores on a scale
  Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Week 8, n=1238,1187 | 0.42 (0.169) | 0.78 (0.172)
  Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Week 12, n=1237,1227 | 0.60 (0.171) | 0.71 (0.172)
  Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Week 28, n=968,956 | 0.16 (0.197) | 0.04 (0.198)
  Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Week 52, n=804,780 | -0.32 (0.218) | -0.12 (0.221)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9320, MMRM; LS mean difference = -0.36, 95% CI 2-sided [-0.83 to 0.11] — Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time,current ESA use at randomization, region,Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6761, MMRM; LS mean difference = -0.11, 95% CI 2-sided [-0.59 to 0.36] — Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented,with factors for treatment, time,current ESA use at randomization, region, Baseline value and Baseline value by time & treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3335, MMRM; LS mean difference = 0.12, 95% CI 2-sided [-0.43 to 0.67] — Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented,with factors for treatment, time,current ESA use at randomization, region, Baseline value and Baseline value by time & treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7423, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.81 to 0.41] — Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented,with factors for treatment, time,current ESA use at randomization, region, Baseline value and Baseline value by time & treatment by time interactions

33. Secondary Outcome: Change From Baseline in On-treatment Mental Component Score (MCS) Using SF-36 HRQoL Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). MCS is an average score derived from 4 domains (vitality, social functioning, role-emotional and mental health) representing overall mental health. MCS ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1238 | 1227
Scores on a scale
  Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Week 8, n=1238,1187 | 0.08 (0.217) | 0.37 (0.221)
  Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Week 12, n=1237,1227 | 0.02 (0.223) | 0.18 (0.224)
  Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Week 28, n=968,956 | -0.35 (0.244) | -0.02 (0.245)
  Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Week 52, n=804,780 | -0.71 (0.290) | -0.35 (0.294)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8268, MMRM; LS mean difference = -0.29, 95% CI 2-sided [-0.90 to 0.32] — Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented,with factors for treatment, time,current ESA use at randomization, region, Baseline value and Baseline value by time & treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6851, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.77 to 0.47] — [estimate comment as in outcome 32, analysis 2]
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8316, MMRM; LS mean difference = -0.33, 95% CI 2-sided [-1.01 to 0.35] — [estimate comment as in outcome 32, analysis 3]
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8032, MMRM; LS mean difference = -0.35, 95% CI 2-sided [-1.16 to 0.46] — [estimate comment as in outcome 32, analysis 4]

34. Secondary Outcome: Change From Baseline in On-treatment SF-36 HRQoL Scores for Bodily Pain, General Health, Mental Health, Role-Emotional, Role-Physical, Social Functioning at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: bodily pain (b pain), general health (GH), mental health (MH), role-emotional (RE) (role limitations caused by emotional problems), role-physical (RP) (role limitations caused by physical problems), social functioning (SF), physical functioning and vitality. Each domain is scored from 0 (poorer health) to 100 (better health). Each domain score ranges from 0 to 100, higher score indicates a better health state and better functioning. Change from Baseline (BL) was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1238 | 1227
Scores on a scale
  Bodily pain: Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Bodily pain: Week 8, n=1238,1187 | 0.11 (0.221) | 0.45 (0.225)
  Bodily pain: Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Bodily pain: Week 12, n=1237,1227 | 0.35 (0.223) | 0.50 (0.224)
  Bodily pain: Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Bodily pain: Week 28, n=968,956 | -0.48 (0.261) | 0.02 (0.263)
  Bodily pain: Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Bodily pain: Week 52, n=804,780 | -0.34 (0.283) | 0.13 (0.288)
  General health: Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  General health: Week 8, n=1238,1187 | 0.36 (0.171) | 0.43 (0.174)
  General health: Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  General health: Week 12, n=1237,1227 | 0.28 (0.174) | 0.48 (0.175)
  General health: Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  General health: Week 28, n=968,956 | 0.14 (0.200) | 0.04 (0.201)
  General health: Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  General health: Week 52, n=804,780 | -0.27 (0.220) | -0.19 (0.224)
  Mental health: Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Mental health: Week 8, n=1238,1187 | -0.19 (0.204) | 0.12 (0.208)
  Mental health: Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Mental health: Week 12, n=1237,1227 | -0.07 (0.210) | -0.09 (0.211)
  Mental health: Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Mental health: Week 28, n=968,956 | -0.67 (0.231) | -0.37 (0.232)
  Mental health: Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Mental health: Week 52, n=804,780 | -0.85 (0.271) | -0.61 (0.275)
  Role-emotional: Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Role-emotional: Week 8, n=1238,1187 | 0.45 (0.253) | 0.54 (0.258)
  Role-emotional: Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Role-emotional: Week 12, n=1237,1227 | 0.17 (0.258) | 0.43 (0.259)
  Role-emotional: Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Role-emotional: Week 28, n=968,956 | -0.30 (0.290) | 0.07 (0.292)
  Role-emotional: Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Role-emotional: Week 52, n=804,780 | -0.90 (0.339) | -0.38 (0.344)
  Role-physical: Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Role-physical: Week 8, n=1238,1187 | 0.33 (0.202) | 0.83 (0.205)
  Role-physical: Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Role-physical: Week 12, n=1237,1227 | 0.40 (0.203) | 0.73 (0.204)
  Role-physical: Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Role-physical: Week 28, n=968,956 | 0.06 (0.230) | 0.00 (0.232)
  Role-physical: Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Role-physical: Week 52, n=804,780 | -0.63 (0.259) | -0.44 (0.263)
  Social functioning: Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Social functioning: Week 8, n=1238,1187 | 0.19 (0.224) | 0.82 (0.228)
  Social functioning: Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Social functioning: Week 12, n=1237,1227 | 0.21 (0.224) | 0.53 (0.225)
  Social functioning: Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Social functioning: Week 28, n=968,956 | 0.04 (0.247) | 0.17 (0.249)
  Social functioning: Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Social functioning: Week 52, n=804,780 | -0.58 (0.282) | -0.20 (0.286)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8562, MMRM; LS mean difference = -0.34, 95% CI 2-sided [-0.95 to 0.28] — B pain,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6849, MMRM; LS mean difference = -0.15, 95% CI 2-sided [-0.77 to 0.47] — B pain,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9074, MMRM; LS mean difference = -0.49, 95% CI 2-sided [-1.22 to 0.24] — B pain,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8765, MMRM; LS mean difference = -0.47, 95% CI 2-sided [-1.26 to 0.32] — B pain,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 5: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6252, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.56 to 0.40] — GH,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 6: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7852, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.68 to 0.29] — GH,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 7: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3614, MMRM; LS mean difference = 0.10, 95% CI 2-sided [-0.46 to 0.66] — GH,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 8: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5991, MMRM; LS mean difference = -0.08, 95% CI 2-sided [-0.70 to 0.54] — GH,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 9: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8526, MMRM; LS mean difference = -0.31, 95% CI 2-sided [-0.88 to 0.27] — MH,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 10: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.4673, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.56 to 0.61] — MH,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 11: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8262, MMRM; LS mean difference = -0.31, 95% CI 2-sided [-0.95 to 0.33] — MH,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 12: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7380, MMRM; LS mean difference = -0.25, 95% CI 2-sided [-1.00 to 0.51] — MH,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 13: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5997, MMRM; LS mean difference = -0.09, 95% CI 2-sided [-0.80 to 0.62] — RE,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 14: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7649, MMRM; LS mean difference = -0.26, 95% CI 2-sided [-0.98 to 0.45] — RE,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 15: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8175, MMRM; LS mean difference = -0.37, 95% CI 2-sided [-1.18 to 0.43] — RE,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 16: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8591, MMRM; LS mean difference = -0.52, 95% CI 2-sided [-1.47 to 0.43] — RE,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 17: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9588, MMRM; LS mean difference = -0.50, 95% CI 2-sided [-1.06 to 0.06] — RP,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 18: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8761, MMRM; LS mean difference = -0.33, 95% CI 2-sided [-0.90 to 0.23] — RP,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 19: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.4293, MMRM; LS mean difference = 0.06, 95% CI 2-sided [-0.58 to 0.70] — RP,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 20: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6983, MMRM; LS mean difference = -0.19, 95% CI 2-sided [-0.92 to 0.53] — RP,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 21: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9743, MMRM; LS mean difference = -0.62, 95% CI 2-sided [-1.25 to 0.00] — SF,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 22: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8405, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-0.94 to 0.31] — SF,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time,current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 23: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6459, MMRM; LS mean difference = -0.13, 95% CI 2-sided [-0.82 to 0.56] — SF,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 24: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8272, MMRM; LS mean difference = -0.38, 95% CI 2-sided [-1.17 to 0.41] — SF,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions

35. Secondary Outcome: Change From Baseline in On-treatment Vitality Scores Using SF-36 HRQoL Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). Vitality score ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1238 | 1227
Scores on a scale
  Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Week 8, n=1238,1187 | 0.35 (0.192) | 0.90 (0.195)
  Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Week 12, n=1237,1227 | 0.62 (0.200) | 0.74 (0.201)
  Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Week 28, n=968,956 | 0.22 (0.222) | 0.32 (0.223)
  Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Week 52, n=804,780 | -0.14 (0.250) | 0.35 (0.253)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9786, MMRM; LS mean difference = -0.56, 95% CI 2-sided [-1.09 to -0.02] — Week 8: Model was fitted from Baseline up to Week 52 and model adjusted Week 8 data has been presented,with factors for treatment, time,current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6642, MMRM; LS mean difference = -0.12, 95% CI 2-sided [-0.68 to 0.44] — Week 12: Model was fitted from Baseline up to Week 52 and model adjusted Week 12 data has been presented,with factors for treatment, time,current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6261, MMRM; LS mean difference = -0.10, 95% CI 2-sided [-0.72 to 0.52] — Week 28: Model was fitted from Baseline up to Week 52 and model adjusted Week 28 data has been presented,with factors for treatment, time,current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9161, MMRM; LS mean difference = -0.49, 95% CI 2-sided [-1.19 to 0.21] — Week 52: Model was fitted from Baseline up to Week 52 and model adjusted Week 52 data has been presented,with factors for treatment, time,current ESA use at randomization, region, BL value and BL value by time & treatment by time interactions

36. Secondary Outcome: Change From Baseline in On-treatment Physical Functioning Domain Scores Using SF-36 HRQoL Questionnaire at Weeks 8, 12, 28, 52
Description: The SF-36 acute version 2 is a 36-item generic quality of life instrument designed to measure a participant's level of performance in the following 8 health domains: physical functioning, role-physical (role limitations caused by physical problems), social functioning, bodily pain, mental health, role-emotional (role limitations caused by emotional problems), vitality and general health. Each domain is scored from 0 (poorer health) to 100 (better health). Physical functioning score ranges from 0 to 100; higher scores represent better health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1238 | 1227
Scores on a scale
  Week 8, n=1238,1187: number analyzed (Participants) | 1238 | 1187
  Week 8, n=1238,1187 | 0.51 (0.200) | 0.83 (0.203)
  Week 12, n=1237,1227: number analyzed (Participants) | 1237 | 1227
  Week 12, n=1237,1227 | 0.65 (0.195) | 0.52 (0.196)
  Week 28, n=968,956: number analyzed (Participants) | 968 | 956
  Week 28, n=968,956 | 0.05 (0.224) | -0.10 (0.225)
  Week 52, n=804,780: number analyzed (Participants) | 804 | 780
  Week 52, n=804,780 | -0.69 (0.262) | -0.37 (0.266)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8703, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-0.88 to 0.24] — [estimate comment as in outcome 35, analysis 1]
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3167, MMRM; LS mean difference = 0.13, 95% CI 2-sided [-0.41 to 0.67] — [estimate comment as in outcome 35, analysis 2]
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3155, MMRM; LS mean difference = 0.15, 95% CI 2-sided [-0.47 to 0.78] — [estimate comment as in outcome 35, analysis 3]
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8069, MMRM; LS mean difference = -0.32, 95% CI 2-sided [-1.06 to 0.41] — [estimate comment as in outcome 35, analysis 4]

37. Secondary Outcome: Change From Baseline in On-treatment Health Utility EuroQol 5 Dimensions 5 Level (EQ-5D-5L) Questionnaire Score at Week 52
Description: EQ-5D-5L is self-assessment questionnaire, consisting of 5 items covering 5 dimensions (mobility, self care, usual activities, pain/discomfort and anxiety/depression). Each dimension is measured by 5-point Likert scale (1=no problems, 2=slight problems, 3=moderate problems, 4=severe problems and 5=extreme problems). Responses for 5 dimensions together formed a 5-figure description of health state (e.g.11111 indicates no problems in all 5 dimensions). Each of these 5 figure health states were converted to a single index score by applying country-specific value set formula that attaches weights to dimensions and levels. Range for EQ-5D-5L index score is -0.594 (worst health) to 1 (full health state). Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was latest non-missing pre-dose assessment on or before randomization date.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 443 | 399
Scores on a scale | -0.0253 (0.00842) | -0.0018 (0.00883)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9724, MMRM; LS mean difference = -0.0234, 95% CI 2-sided [-0.0474 to 0.0005] — MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, current ESA use, region, Baseline value and Baseline value by time and treatment by time interactions

38. Secondary Outcome: Change From Baseline in On-treatment EQ Visual Analogue Scale (EQ-VAS) at Week 52
Description: The EQ VAS records the respondent's self-rated health on a vertical VAS, ranging from 0 to 100, where 0 represents the worst imaginable health and 100 represents the best imaginable health. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 443 | 399
Scores on a scale | -0.7 (0.78) | -1.4 (0.82)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.2687, MMRM; LS mean difference = 0.7, 95% CI 2-sided [-1.5 to 2.9] — [estimate comment as in outcome 37, analysis 1]

39. Secondary Outcome: Change From Baseline in On-treatment Chronic Kidney Disease- Anemia Symptoms Questionnaire (CKD-AQ) at Weeks 8, 12, 28, 52
Description: CKD-AQ is 21-item patient reported outcome measure assessing symptoms and symptom impact in participants with anemia associated with CKD. It had 3 domains: 1.Tired/Low Energy (LE)/Weak scale consisting of 10 items; 2.Chest Pain (CP)/Shortness of Breath (SOB) scale consisting of 4 items; and 3.Cognitive (Cog) scale consisting of 3 items. The 4 CKD-AQ single items are: shortness of breath, no activity; severity-short breath (S-SB), resting; difficulty standing (diff. std.)for long time (LT) and difficulty sleeping (diff sleep). Single-item were recorded based on a 0-100 scoring with 0=worst possible and 100=best possible score. Three domains scores were calculated as average of items in each domain and ranged from 0-100 where 0=worst possible and 100=best possible score. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Day 1) and Weeks 8, 12, 28, 52
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1341 | 1360
Scores on a scale
  Tired/Low energy/Weak domain: Week 8,n=1340,1294: number analyzed (Participants) | 1340 | 1294
  Tired/Low energy/Weak domain: Week 8,n=1340,1294 | 1.72 (0.424) | 2.94 (0.429)
  Tired/Low energy/Weak domain: Week 12,n=1341,1360 | 2.11 (0.437) | 3.08 (0.434)
  Tired/Low energy/Weak domain: Week 28,n=1053,1047: number analyzed (Participants) | 1053 | 1047
  Tired/Low energy/Weak domain: Week 28,n=1053,1047 | 1.27 (0.495) | 1.87 (0.496)
  Tired/Low energy/Weak domain: Week 52,n=870,865: number analyzed (Participants) | 870 | 865
  Tired/Low energy/Weak domain: Week 52,n=870,865 | 0.20 (0.554) | 1.77 (0.556)
  Chest pain/SOB domain: Week 8,n=1340,1294: number analyzed (Participants) | 1340 | 1294
  Chest pain/SOB domain: Week 8,n=1340,1294 | 0.63 (0.358) | 1.83 (0.363)
  Chest pain/ SOB domain: Week 12,n=1341,1360 | 0.88 (0.370) | 1.53 (0.368)
  Chest pain/ SOB domain: Week 28,n=1053,1047: number analyzed (Participants) | 1053 | 1047
  Chest pain/ SOB domain: Week 28,n=1053,1047 | 0.01 (0.424) | 0.53 (0.425)
  Chest pain/ SOB domain: Week 52,n=870,865: number analyzed (Participants) | 870 | 865
  Chest pain/ SOB domain: Week 52,n=870,865 | -0.71 (0.471) | 0.47 (0.473)
  Cognitive domain: Week 8,n=1340,1294: number analyzed (Participants) | 1340 | 1294
  Cognitive domain: Week 8,n=1340,1294 | 0.13 (0.413) | 0.89 (0.419)
  Cognitive domain: Week 12,n=1341,1360 | -0.17 (0.414) | 1.01 (0.412)
  Cognitive domain: Week 28,n=1053,1047: number analyzed (Participants) | 1053 | 1047
  Cognitive domain: Week 28,n=1053,1047 | -0.40 (0.468) | 0.37 (0.469)
  Cognitive domain: Week 52,n=870,865: number analyzed (Participants) | 870 | 865
  Cognitive domain: Week 52,n=870,865 | -2.00 (0.526) | -0.35 (0.527)
  SOB, no activity: Week 8,n=1340,1294: number analyzed (Participants) | 1340 | 1294
  SOB, no activity: Week 8,n=1340,1294 | -0.1 (0.42) | 1.0 (0.42)
  SOB, no activity: Week 12,n=1341,1360 | 0.1 (0.43) | 0.4 (0.42)
  SOB, no activity: Week 28,n=1053,1047: number analyzed (Participants) | 1053 | 1047
  SOB, no activity: Week 28,n=1053,1047 | -1.1 (0.50) | -0.2 (0.50)
  SOB, no activity: Week 52,n=870,865: number analyzed (Participants) | 870 | 865
  SOB, no activity: Week 52,n=870,865 | -1.7 (0.57) | -1.6 (0.57)
  Severity-short breath, Resting: Week 8,n=1340,1294: number analyzed (Participants) | 1340 | 1294
  Severity-short breath, Resting: Week 8,n=1340,1294 | -0.3 (0.40) | 0.8 (0.40)
  Severity-short breath, Resting:Week 12,n=1341,1360 | -0.3 (0.42) | 0.0 (0.42)
  Severity-short breath, Resting:Week 28,n=1053,1047: number analyzed (Participants) | 1053 | 1047
  Severity-short breath, Resting:Week 28,n=1053,1047 | -1.1 (0.48) | -0.7 (0.48)
  Severity-short breath, Resting:Week 52,n=870,865: number analyzed (Participants) | 870 | 865
  Severity-short breath, Resting:Week 52,n=870,865 | -2.0 (0.53) | -0.5 (0.53)
  Diff std for long time: Week 8,n=1340,1294: number analyzed (Participants) | 1340 | 1294
  Diff std for long time: Week 8,n=1340,1294 | 1.0 (0.62) | 2.5 (0.63)
  Diff std for long time: Week 12,n=1341,1360 | 0.7 (0.63) | 1.6 (0.62)
  Diff std for long time: Week 28,n=1053,1047: number analyzed (Participants) | 1053 | 1047
  Diff std for long time: Week 28,n=1053,1047 | 0.4 (0.71) | 1.7 (0.71)
  Diff std for long time: Week 52,n=870,865: number analyzed (Participants) | 870 | 865
  Diff std for long time: Week 52,n=870,865 | -2.1 (0.76) | 1.2 (0.76)
  Difficulty sleeping: Week 8,n=1340,1294: number analyzed (Participants) | 1340 | 1294
  Difficulty sleeping: Week 8,n=1340,1294 | 1.6 (0.60) | 1.1 (0.61)
  Difficulty sleeping: Week 12,n=1341,1360 | 0.5 (0.60) | 2.0 (0.59)
  Difficulty sleeping: Week 28,n=1053,1047: number analyzed (Participants) | 1053 | 1047
  Difficulty sleeping: Week 28,n=1053,1047 | -0.7 (0.69) | -0.3 (0.70)
  Difficulty sleeping: Week 52,n=870,865: number analyzed (Participants) | 870 | 865
  Difficulty sleeping: Week 52,n=870,865 | -2.6 (0.78) | -0.3 (0.78)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9780, MMRM; LS mean difference = -1.22, 95% CI 2-sided [-2.40 to -0.03] — Tired/LE/Weak domain,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9430, MMRM; LS mean difference = -0.97, 95% CI 2-sided [-2.18 to 0.23] — Tired/LE/Weak domain,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8042, MMRM; LS mean difference = -0.60, 95% CI 2-sided [-1.98 to 0.77] — Tired/LE/Weak domain,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9770, MMRM; LS mean difference = -1.57, 95% CI 2-sided [-3.11 to -0.03] — Tired/LE/Weak domain,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 5: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9905, MMRM; LS mean difference = -1.20, 95% CI 2-sided [-2.20 to -0.20] — CP/SOB,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 6: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8939, LS mean difference; LS mean difference = -0.65, 95% CI 2-sided [-1.67 to 0.37] — CP/SOB,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 7: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8070, MMRM; LS mean difference = -0.52, 95% CI 2-sided [-1.70 to 0.66] — CP/SOB,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 8: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9615, MMRM; LS mean difference = -1.18, 95% CI 2-sided [-2.49 to 0.13] — CP/SOB,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 9: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9015, MMRM; LS mean difference = -0.76, 95% CI 2-sided [-1.91 to 0.39] — Cog domain,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 10: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9781, MMRM; LS mean difference = -1.18, 95% CI 2-sided [-2.32 to -0.03] — Cog domain,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 11: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8778, MMRM; LS mean difference = -0.77, 95% CI 2-sided [-2.07 to 0.53] — Cog domain,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 12: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9864, MMRM; LS mean difference = -1.65, 95% CI 2-sided [-3.11 to -0.19] — Cog domain,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 13: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9725, MMRM; LS mean difference = -1.1, 95% CI 2-sided [-2.3 to 0.0] — SOB, no activity,Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 14: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7188, MMRM; LS mean difference = -0.3, 95% CI 2-sided [-1.5 to 0.8] — SOB, no activity,Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 15: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8903, MMRM; LS mean difference = -0.9, 95% CI 2-sided [-2.3 to 0.5] — SOB, no activity,Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 16: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.5011, MMRM; LS mean difference = 0.0, 95% CI 2-sided [-1.6 to 1.6] — SOB, no activity,Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 17: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9716, MMRM; LS mean difference = -1.1, 95% CI 2-sided [-2.2 to 0.0] — S-SB,Resting, Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 18: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6908, MMRM; LS mean difference = -0.3, 95% CI 2-sided [-1.4 to 0.9] — S-SB,Resting, Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 19: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7462, MMRM; LS mean difference = -0.5, 95% CI 2-sided [-1.8 to 0.9] — S-SB,Resting, Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 20: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9770, MMRM; LS mean difference = -1.5, 95% CI 2-sided [-2.9 to 0.0] — S-SB,Resting, Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 21: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9471, MMRM; LS mean difference = -1.4, 95% CI 2-sided [-3.2 to 0.3] — Diff std for LT, Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 22: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8330, MMRM; LS mean difference = -0.9, 95% CI 2-sided [-2.6 to 0.9] — Diff std for LT, Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 23: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8918, MMRM; LS mean difference = -1.2, 95% CI 2-sided [-3.2 to 0.7] — Diff std for LT, Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 24: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9986, MMRM; LS mean difference = -3.2, 95% CI 2-sided [-5.4 to -1.1] — Diff std for LT, Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 25: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.3035, MMRM; LS mean difference = 0.4, 95% CI 2-sided [-1.2 to 2.1] — Diff sleep, Week8:Model was fitted from Baseline up to Week52 and model adjusted Week8 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 26: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9563, MMRM; LS mean difference = -1.4, 95% CI 2-sided [-3.1 to 0.2] — Diff sleep, Week12:Model was fitted from Baseline up to Week52 and model adjusted Week12 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 27: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6548, MMRM; LS mean difference = -0.4, 95% CI 2-sided [-2.3 to 1.5] — Diff sleep, Week28:Model was fitted from Baseline up to Week52 and model adjusted Week28 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions
Statistical Analysis 28: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9832, MMRM; LS mean difference = -2.4, 95% CI 2-sided [-4.5 to -0.2] — Diff sleep, Week52:Model was fitted from Baseline up to Week52 and model adjusted Week52 data has been presented, with factors for treatment, time, current ESA use, region, BL value and BL value by time and treatment by time interactions

40. Secondary Outcome: Change From Baseline in On-treatment Patient Global Impression of Severity (PGI-S) at Weeks 8, 12, 28, 52
Description: The PGI-S is a 1-item questionnaire designed to assess participant's impression of disease severity on a 5-point disease severity scale (0=absent, 1=mild, 2=moderate, 3=severe, or 4=very severe). A higher score indicated more disease severity. Change from Baseline was calculated as on-treatment visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1), Weeks 8, 12, 28 and 52
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1341 | 1362
Scores on a scale
  Week 8, n=1341,1295: number analyzed (Participants) | 1341 | 1295
  Week 8, n=1341,1295 | 0.00 (0.022) | -0.02 (0.022)
  Week 12, n=1341,1362 | 0.03 (0.022) | -0.02 (0.022)
  Week 28, n=1054,1051: number analyzed (Participants) | 1054 | 1051
  Week 28, n=1054,1051 | 0.05 (0.025) | 0.09 (0.025)
  Week 52, n=871,865: number analyzed (Participants) | 871 | 865
  Week 52, n=871,865 | 0.11 (0.028) | 0.06 (0.029)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.6917, MMRM; LS mean difference = 0.02, 95% CI 2-sided [-0.05 to 0.08] — Week 8: Model was fitted from Baseline up to Week52 and model adjusted Week 8 data has been presented, with factors for treatment, time, current ESA use, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 2: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.9510, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.01 to 0.11] — Week 12: Model was fitted from Baseline up to Week52 and model adjusted Week 12 data has been presented, with factors for treatment, time, current ESA use, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 3: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.1136, MMRM; LS mean difference = -0.04, 95% CI 2-sided [-0.11 to 0.03] — Week 28: Model was fitted from Baseline up to Week52 and model adjusted Week 28 data has been presented, with factors for treatment, time, current ESA use, region, Baseline value and Baseline value by time and treatment by time interactions
Statistical Analysis 4: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.8859, MMRM; LS mean difference = 0.05, 95% CI 2-sided [-0.03 to 0.13] — Week 52: Model was fitted from Baseline up to Week52 and model adjusted Week 52 data has been presented, with factors for treatment, time, current ESA use, region, Baseline value and Baseline value by time and treatment by time interactions

41. Secondary Outcome: Change From Baseline in Post-randomization Estimated Glomerular Filtration Rate (eGFR) at Week 52
Description: Blood samples were collected to analyze estimated glomerular filtration rate. Change from Baseline was calculated as post-Baseline visit value minus Baseline value. Baseline was defined as the latest non-missing pre-dose assessment on or before the randomization date.
Time Frame: Baseline (Pre-dose on Day 1) and Week 52
Population: All Randomized (ITT) Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mL per minute per 1.73 square meter
Arm/Group | Daprodustat | Darbepoetin Alfa
Number analyzed (Participants) | 1869 | 1868
mL per minute per 1.73 square meter | -2.88 (0.193) | -2.67 (0.193)
Statistical Analysis 1: Comparison: Daprodustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.7716, MMRM; LS mean difference = -0.20, 95% CI 2-sided [-0.74 to 0.33] — MMRM model was fitted from Baseline up to Week 52 with factors for treatment, time, current ESA use at randomization, region, Baseline value and Baseline value by time and treatment by time interactions

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-SAEs were collected from Week -4 up to randomization (Day 1) during Run-in placebo period. All-cause mortality, treatment emergent serious adverse events (TESAEs) and non-serious treatment emergent adverse events (non-STEAEs) were collected from randomization (Day 1) up to 4.3 person-years for CV follow-up time period (Treatment Period)
Description: All-cause mortality and Placebo run-in(SAEs/Non-SAEs)used All Randomized(ITT)Population consisting of all randomized participants and analyzed based on treatment to which they were randomized.TESAEs/non-serious TEAEs during treatment period used Safety Population, included all randomized participants who received at least 1 dose of treatment and analyzed based on treatment received.2 participants in All Randomized(ITT)Population did not receive treatment and were excluded from Safety Population.
Groups:
- Run-in Period: Placebo: Participants received placebo tablets orally once daily in run-in period from Week-4 up to randomization (Day 1).
- Daprodustat: Participants received treatment with daprodustat film-coated tablets at dose levels ranging from 1, 2, 4, 6, 8, 10, 12, 16 and 24 milligrams (mg) orally once daily from randomization (Day 1) up to 51.1 month. Study treatment was dose-titrated to achieve and maintain hemoglobin (Hgb) in the target range (10 to 11 grams per deciliter [g/dL]).
- Darbepoetin Alfa: Participants received treatment with darbepoetin alfa as prefilled syringes (PFS) for subcutaneous or intravenous (IV) injection at 4-weekly total dose levels ranging from 20, 30, 40, 60, 80, 100, 150, 200, 300 and 400 microgram (mcg) from randomization (Day 1) up to 51.1 month. Darbepoetin alfa IV injection was administered to participants undergoing hemodialysis. Study treatment was dose-titrated to achieve and maintain Hgb in the target range (10 to 11 g/dL).
Arm/Group | Run-in Period: Placebo | Daprodustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 0/3872 | 301/1937 | 298/1935
Serious Adverse Events (participants affected / at risk) | 63/3872 | 850/1937 | 703/1933
Other Adverse Events (participants affected / at risk) | 0/3872 | 851/1937 | 825/1933
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Run-in Period: Placebo (N=3872) | Daprodustat (N=1937) | Darbepoetin Alfa (N=1933)
Pneumonia (Infections and infestations) | 3 (3) | 78 (90) | 75 (81)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 86 (90) | 49 (52)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 70 (76) | 47 (53)
Azotaemia (Renal and urinary disorders) | 1 (1) | 54 (56) | 35 (35)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 48 (50) | 36 (37)
COVID-19 (Infections and infestations) | 1 (1) | 39 (39) | 33 (33)
Urinary tract infection (Infections and infestations) | 2 (2) | 33 (34) | 36 (38)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 33 (34) | 31 (34)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 37 (40) | 26 (28)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 26 (26) | 25 (26)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 29 (43) | 20 (23)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 25 (27) | 23 (24)
Cardiac failure (Cardiac disorders) | 2 (2) | 28 (35) | 14 (17)
Cellulitis (Infections and infestations) | 3 (3) | 19 (22) | 14 (15)
Sepsis (Infections and infestations) | 0 (0) | 14 (15) | 19 (19)
Peritonitis (Infections and infestations) | 0 (0) | 21 (28) | 10 (15)
Renal impairment (Renal and urinary disorders) | 0 (0) | 20 (21) | 11 (11)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 16 (20) | 13 (16)
Angina unstable (Cardiac disorders) | 0 (0) | 13 (15) | 15 (17)
Hypertension (Vascular disorders) | 1 (1) | 15 (16) | 11 (14)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 10 (12) | 16 (20)
Renal failure (Renal and urinary disorders) | 0 (0) | 15 (16) | 11 (11)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 11 (11) | 11 (13)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 13 (13) | 8 (8)
Coronary artery disease (Cardiac disorders) | 0 (0) | 10 (12) | 11 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 13 (14) | 7 (7)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 8 (8) | 12 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (10) | 11 (12)
Angina pectoris (Cardiac disorders) | 0 (0) | 10 (10) | 9 (9)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 11 (12) | 8 (9)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 12 (13) | 7 (7)
Device malfunction (Product Issues) | 0 (0) | 9 (10) | 9 (12)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 12 (12) | 6 (6)
Death (General disorders) | 0 (0) | 13 (13) | 4 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 7 (8) | 10 (10)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 7 (7) | 10 (11)
Myocardial infarction (Cardiac disorders) | 0 (0) | 14 (14) | 3 (3)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 12 (14)
Hypertensive crisis (Vascular disorders) | 1 (1) | 8 (10) | 8 (8)
Hypertensive urgency (Vascular disorders) | 0 (0) | 7 (10) | 9 (9)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 9 (9) | 6 (6)
Hypotension (Vascular disorders) | 0 (0) | 10 (10) | 5 (5)
Non-cardiac chest pain (General disorders) | 0 (0) | 9 (9) | 6 (8)
Osteomyelitis (Infections and infestations) | 0 (0) | 7 (10) | 8 (9)
Syncope (Nervous system disorders) | 0 (0) | 6 (6) | 9 (9)
Urosepsis (Infections and infestations) | 0 (0) | 5 (5) | 10 (10)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 9 (10)
Cardiac arrest (Cardiac disorders) | 0 (0) | 10 (10) | 4 (4)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 9 (12) | 5 (5)
Device related infection (Infections and infestations) | 0 (0) | 7 (8) | 7 (10)
Gangrene (Infections and infestations) | 0 (0) | 8 (8) | 6 (8)
Hypertensive emergency (Vascular disorders) | 2 (2) | 6 (8) | 8 (8)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 12 (14) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 7 (7) | 6 (6)
Device related sepsis (Infections and infestations) | 0 (0) | 7 (8) | 5 (5)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 7 (8) | 5 (7)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 7 (7) | 5 (5)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 7 (9) | 5 (5)
Nephropathy (Renal and urinary disorders) | 0 (0) | 6 (6) | 6 (6)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 4 (4) | 8 (8)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 7 (7)
Bronchitis (Infections and infestations) | 1 (1) | 4 (4) | 7 (7)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (8) | 5 (5)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 6 (6) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 7 (7) | 4 (4)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 6 (6) | 4 (4)
Bradycardia (Cardiac disorders) | 1 (1) | 7 (7) | 3 (3)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 7 (9) | 3 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4) | 6 (6)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 5 (5) | 5 (5)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 6 (6) | 4 (4)
Pyelonephritis (Infections and infestations) | 0 (0) | 3 (3) | 7 (7)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 7 (7) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 4 (4) | 6 (6)
Gastritis (Gastrointestinal disorders) | 1 (1) | 4 (4) | 5 (5)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 7 (7) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 5 (5) | 4 (6)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 6 (6) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 5 (6)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 5 (5)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 7 (7) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 4 (4) | 4 (4)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 6 (6) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 2 (2)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 4 (4)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 2 (3)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 5 (5) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 4 (5)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (9)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 6 (8) | 1 (3)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 3 (3) | 4 (4)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 4 (4) | 3 (4)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 6 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 6 (7)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 5 (5)
Aortic stenosis (Vascular disorders) | 0 (0) | 5 (5) | 1 (1)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 (0) | 6 (7) | 0 (0)
Chest pain (General disorders) | 1 (1) | 4 (5) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Generalised oedema (General disorders) | 0 (0) | 2 (3) | 4 (4)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 3 (3)
Influenza (Infections and infestations) | 0 (0) | 5 (5) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 2 (3)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 5 (6) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2) | 4 (4)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 3 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3)
Pyrexia (General disorders) | 1 (1) | 2 (2) | 4 (4)
Seizure (Nervous system disorders) | 0 (0) | 4 (4) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 3 (4) | 3 (3)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 3 (3)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 4 (6)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0)
Blood creatinine increased (Investigations) | 2 (2) | 4 (4) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 4 (4) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2)
Cerebral infarction (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1)
Device occlusion (Product Issues) | 0 (0) | 4 (4) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Haematoma (Vascular disorders) | 0 (0) | 3 (3) | 2 (2)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 3 (3) | 2 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 3 (3) | 2 (2)
Post procedural infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 2 (3) | 3 (3)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 4 (4)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 4 (4)
Arteriovenous fistula site infection (Infections and infestations) | 0 (0) | 2 (3) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Asthenia (General disorders) | 1 (1) | 3 (3) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 3 (3) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (4)
Haematuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 2 (3)
Intermittent claudication (Vascular disorders) | 0 (0) | 3 (3) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 2 (2)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1) | 3 (4)
Pericardial effusion (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3)
Renal cyst haemorrhage (Renal and urinary disorders) | 0 (0) | 2 (2) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 3 (4)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 3 (3) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 3 (3) | 1 (2)
Acute hepatitis B (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Catheter site infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Endocarditis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Endophthalmitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (3) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Haemodialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 2 (2)
Nephropathy toxic (Renal and urinary disorders) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 1 (1)
Pericarditis uraemic (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (3)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 2 (4)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebellar stroke (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Dementia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 2 (2)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Diabetic gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Dialysis hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Diastolic dysfunction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Enterococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Fungal peritonitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 2 (2)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Intercostal neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Intracranial haematoma (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Ischaemic skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Melaena (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Peritonitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Renal transplant failure (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Retinal detachment (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 2 (2)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Uraemic gastropathy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Acid base balance abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Acute abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Anuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Aortic intramural haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Arteriovenous fistula site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft site infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Basilar artery occlusion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood loss anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Brain stem infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site extravasation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Coagulation test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (2)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Complication associated with device (General disorders) | 0 (0) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Congestive cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cryptogenic cirrhosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Cutaneous calcification (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cystitis klebsiella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dengue haemorrhagic fever (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Device failure (Product Issues) | 0 (0) | 1 (1) | 0 (0)
Diabetic end stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic gastropathy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidotic hyperglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis intestinal haemorrhagic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Duodenitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dystonic tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram QRS complex prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1)
Embolic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Emphysematous pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Endometrial cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Erythrodermic psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Evans syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Gait inability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis Escherichia coli (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis bacillus (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Giant cell arteritis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Gliosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Glomerulonephritis chronic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Glomerulonephritis membranous (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Gouty tophus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematological malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemobilia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Heart injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Hepatic cyst infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes ophthalmic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (3)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperprolactinaemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemic syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
IIIrd nerve paresis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Immobile (Social circumstances) | 0 (0) | 1 (1) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Incision site abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infected fistula (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infective tenosynovitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Intercapillary glomerulosclerosis (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Internal haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intracranial aneurysm (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Kidney transplant rejection (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lead dislodgement (Product Issues) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lumbosacral radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lupus nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm of unknown primary site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolic syndrome (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Necrobiosis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Nerve root injury lumbar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Non-immune heparin associated thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatic enzymes increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Parathyroid hyperplasia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Peau d'orange (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic mass (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia adenoviral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia escherichia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pseudohyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary hypertensive crisis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Putamen haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pyonephrosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Refeeding syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Refractory anaemia with an excess of blasts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cyst infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Renal graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0/0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Right ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (2)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Sarcopenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scrotal swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Serratia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sideroblastic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinusitis fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Sphingomonas paucimobilis infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Starvation ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subclavian artery stenosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Syringomyelia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ulcerative keratitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ureteric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Ureteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular device occlusion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vascular graft complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Vascular graft infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Vertigo CNS origin (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (2)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vitreoretinal traction syndrome (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound secretion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bifascicular block (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Renal artery occlusion (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Period: Placebo (N=3872) | Daprodustat (N=1937) | Darbepoetin Alfa (N=1933)
Hypertension (Vascular disorders) | 0 (0) | 247 (317) | 264 (339)
Oedema peripheral (General disorders) | 0 (0) | 198 (239) | 162 (199)
Urinary tract infection (Infections and infestations) | 0 (0) | 164 (245) | 153 (199)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 149 (181) | 139 (172)
Nasopharyngitis (Infections and infestations) | 0 (0) | 118 (163) | 133 (180)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 128 (148) | 122 (141)
Constipation (Gastrointestinal disorders) | 0 (0) | 127 (150) | 88 (96)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 104 (128) | 88 (119)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 82 (95) | 105 (110)
Nausea (Gastrointestinal disorders) | 0 (0) | 103 (120) | 84 (101)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/35/NCT02876835/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/35/NCT02876835/SAP_001.pdf